CLINICAL TRIAL: NCT05760898
Title: Improving Hypertension Control for Patients With Rheumatoid Arthritis
Brief Title: Improving Hypertension Control in Rheumatoid Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00112307; 3U54MD012530-05S2 (NIH)
Record Dates: First submitted 2023-02-09; First posted 2023-03-09 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-08

CONDITIONS: Hypertension; Rheumatoid Arthritis
MeSH Terms: conditions — Hypertension; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood pressure intervention arm (Experimental): The investigators will recruit 25 RA patients with HTN for the study. Participants will be provided with a home blood pressure monitor, teaching from nursing staff regarding the correct use of the monitor, and a guide to help interpret normal and elevated blood pressure values. Participants will be instructed to obtain and record blood pressure values at least three times per week over the course of 3 months. Every 2 weeks, these results will be sent to the study team, and participants will complete a brief survey regarding other factors that may influence blood pressure control, including RA disease activity (RAPID3 score), pain, current use of acute RA therapies, anti-hypertensive medication use, anti-hypertensive medication adherence, and current perceived barriers to HTN self-management.
  Interventions: Behavioral: Blood pressure intervention arm

INTERVENTIONS:
Behavioral: Blood pressure intervention arm — The intervention will focus on empowering patients to actively participate in their HTN care, facilitating patient-provider communication, and creating a cohesive care team to close the coordination loop for HTN management. This pilot intervention will help achieve these goals by providing participants with home blood pressure monitors and teaching, improving patient-provider communication regarding blood pressure and RA management, and initiating care coordination between rheumatology and primary care providers.

SUMMARY:
Rheumatoid arthritis (RA) is a autoimmune disease associated with an increased risk of developing coronary artery disease (CAD) and premature death,. Traditional CAD risk factors like hypertension (HTN) are both very common and poorly controlled among RA patients. Patients with RA face significant challenges in controlling HTN. The goal of this project is to identify barriers to HTN care in patients with RA to reduce CAD events.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Uncontrolled hypertension
* History of rheumatoid arthritis
* Receive both primary care and rheumatology care from Duke Health System

Exclusion Criteria:

* Age less than 18 years old
* Healthy volunteers without rheumatoid arthritis and hypertension
* Do not receive both primary care and rheumatology care from Duke Health System
* Cognitive impairment with lack the capacity to consent to study participation
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Intervention feasibility as measured by participant accrual rates | 6 months
  Rate at which participants are able to be successfully recruited
Intervention feasibility as measured by participant retention | 6 months
  Percentage of participants who successfully complete the study
Intervention feasibility as measured by adherence to blood pressure monitoring | 6 months
  Percentage of expected blood pressures reported by participants
Intervention feasibility as measured by adherence to survey reporting | 6 months
  Percentage of expected surveys completed by participants
Intervention feasibility as measured by sample characteristics | 6 months
  Description of sociodemographic characteristics of population, rheumatoid arthritis characteristics (eg, duration, medications, severity), and hypertension characteristics (eg, duration, medications, severity)
Intervention feasibility as measured by use of resources | 6 months
  Cost of participant recruitment, education, blood pressure monitors, participant compensation, research coordinator time and cost needed to collect data, and statistical analysis
Intervention feasibility as measured by sustainability of data collection procedures | 6 months
  Financial and time commitments required to successfully collect participant surveys, blood pressure monitoring results, send information to providers, and monitor provider responses
Intervention acceptability as measured by qualitative interviews | 6 months
  Qualitative interviews will be performed at the end of the pilot intervention with all study participants to assess the acceptability of the intervention. Rheumatology and primary care providers caring for study participants will also be invited to comment on the acceptability of the intervention.
Perceived appropriateness of the intervention to address the health care disparity in HTN (hypertension) control for Black RA patients as measured by qualitative interviews | 6 months
  Qualitative interviews will be performed at the end of the pilot intervention with all study participants to assess the perceived appropriateness of the intervention to address the health care disparity in HTN control for Black RA patients. Rheumatology and primary care providers caring for study participants will also be invited to comment on the appropriateness of the intervention.
Barriers to and enablers of participating in the intervention as measured by qualitative interviews | 6 months
  Qualitative interviews will be performed at the end of the pilot intervention with all study participants to assess barriers to and enablers of participating in the intervention.

SECONDARY OUTCOMES:
Participant blood pressure values | 6 months
  Systolic and diastolic blood pressures taken at least three times per week and reported to the study team every 2 weeks for 6 months
Participant rheumatoid arthritis disease activity | 6 months
  Rheumatoid arthritis disease activity self-reported by participants using the RAPID3 score every 2 weeks for 6 months
Participant medication use | 6 months
  Medication use for hypertension and rheumatoid arthritis reported by participants every 2 weeks for 6 months
Anti-hypertensive medication adherence | 6 months
  Participant self-reported adherence percentage to anti-hypertensive medications collected every 2 weeks for 6 months
Perceived barriers to hypertension self-management | 6 months
  Participant self-reported barriers to hypertension self-management collected every 2 weeks for 6 months
Provider engagement as measured by response to study team messages | 6 months
  Frequency and type of provider responses to study team messages
Provider engagement as measured by interactions with participants | 6 months
  Frequency and type of provider interactions with participants after receiving a study team message
Care coordination | 6 months
  Activation of care team members
Number of participants with a change in medical therapy | 6 months
  Changes in anti-hypertensive or RA therapies

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No